CLINICAL TRIAL: NCT04433260
Title: Immediate and Mid-term Implications of the Covid-19 Pandemic on the Physical, Behavioural and Mental Health of Healthcare Workers: A Cohort Study of Doctor, Nurses and Other Health Care Workers
Brief Title: COVID19 and Physical and Emotional Wellbeing of HCP
Acronym: CoPE-HCP
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 284686
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Mental Health
Keywords: healthcare professionals; Personal protective equipment; covid-19; SARS-CoV2
MeSH Terms: conditions — Psychological Well-Being; COVID-19 | interventions — Patient Health Questionnaire; Surveys and Questionnaires; Ethanol; Lead; Informed Consent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cases: Doctors, nurses and other healthcares ≥ 18 years of age in direct contact with patients potentially infected with COVID-19
  Interventions: Other: Questionnaire including validated tools such as Patient Health Questionnaire (PHQ-9), the 7-item Generalised Anxiety Disorder (GAD- 7), the 7-item insomnia severity index; Other: Questionnaire, same tools as before, with inclusion of PCL5 questionnaire too.; Other: Informed consent
- Internal Control: Healthcare /NHS Administrative staff who are working in the hospital, but not directly in contact with patients potentially infected with COVID-19.
  Interventions: Other: Questionnaire including validated tools such as Patient Health Questionnaire (PHQ-9), the 7-item Generalised Anxiety Disorder (GAD- 7), the 7-item insomnia severity index; Other: Questionnaire, same tools as before, with inclusion of PCL5 questionnaire too.; Other: Informed consent
- Population Control: Non-healthcare/non-NHS academic staff who are not working in the environment where patient exposure is expected.
  Interventions: Other: Questionnaire including validated tools such as Patient Health Questionnaire (PHQ-9), the 7-item Generalised Anxiety Disorder (GAD- 7), the 7-item insomnia severity index; Other: Questionnaire, same tools as before, with inclusion of PCL5 questionnaire too.; Other: Informed consent
- Follow-up cases: Doctors, nurses and other healthcare workers ≥ 18 years of age in direct contact with patients potentially infected with COVID-19 consenting to receive follow-up surveys (n ~ 400)
  Interventions: Other: Questionnaire including validated tools such as Patient Health Questionnaire (PHQ-9), the 7-item Generalised Anxiety Disorder (GAD- 7), the 7-item insomnia severity index; Other: Questionnaire, same tools as before, with inclusion of PCL5 questionnaire too.; Other: Informed consent
- Follow-up controls: Healthcare Administrative staff who are working in the hospital, not at risk of work-related exposure to patients potentially infected with COVID-19 (n~80)
  Interventions: Other: Questionnaire including validated tools such as Patient Health Questionnaire (PHQ-9), the 7-item Generalised Anxiety Disorder (GAD- 7), the 7-item insomnia severity index; Other: Questionnaire, same tools as before, with inclusion of PCL5 questionnaire too.; Other: Informed consent

INTERVENTIONS:
Other: Questionnaire including validated tools such as Patient Health Questionnaire (PHQ-9), the 7-item Generalised Anxiety Disorder (GAD- 7), the 7-item insomnia severity index — The electronic survey for phase 1 detailing questions regarding affective symptoms, behaviour and ongoing concerns will be sent and implied consent assumed from responders. A proportion of these patients who give consent to be repeatedly contacted throughout the study period will be recruited into phase 2 of the study at 6 weeks and 4 months
  Other Names: Questionnaire; Questionnaire to evaluate their current quantity and frequency of alcohol use, smoking habit and mental wellbeing score (abbreviated Warwick-Edinburgh).
Other: Questionnaire, same tools as before, with inclusion of PCL5 questionnaire too. — Follow-up electronic surveys including questions regarding affective symptoms, behavioural changes and mental well-being will be sent at 6-weeks and 4-months following the initial survey. This will be sent to participants from Groups 1-3 that provided consent to receive these follow-up questionnaires.
Other: Informed consent — Participants will need to give their consent to participate to the survey after reading PIS

SUMMARY:
The current COVID-19 pandemic has affected more than 3 million people worldwide across more than 200 countries.

In the United Kingdom alone, at the end of April, there were almost 160,000 confirmed cases with more than 20,000 deaths. This has undoubtedly had significant physical and economical impact on the public.

Healthcare workers are at high risk of developing life-threatening infectious diseases with increased exposure to patients' blood and bodily fluids. As such, health care workers arguably experience heightened anxiety and are predisposed to greater negative psycho-social impact from the current COVID-19 pandemic.

The aim of this study is to evaluate the physical and psychological impact of COVID-19 on healthcare workers. This will be performed in two phases.

In phase 1, investigators will collect information to evaluate the current psychiatric symptom profile (in particular, screening for anxiety or depression related symptoms), alcohol use, sleep-related complaints and overall well-being among healthcare workers who participate in this survey (with a focus on junior doctors). In addition the association of these mental health and behavioural parameters with the prevalence of stressful occasions, such as long-hours, unpredictability of work / redeployment, availability of personal protection equipment and concerns regarding family/relationship and self will be assessed.

In phase 2, investigators will then reassess for the development or progression of psychiatric symptoms, use of alcohol and other substances, behavioural or interpersonal relationship changes as well as physical well-being at 6 weeks and 4- months. Physical well-being is assessed through the presence of suspected or confirmed COVID-19 infection and absence from work. Specifically, investigators will study the impact of variable provision of personal protection equipment (supply and training), extended working hours, and concern for well-being of family members, on work morale and anxiety levels.

Another aim is also study the longer term mental health consequences of the current pandemic on health care workers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >=18
2. Electronic consent
3. Either:

a - healthcare workers in contact with patients with confirmed or suspected COVID-19 b - Healthcare staff not having direct patient contact c - Non-healthcare academic staff with no direct patient contact

Exclusion Criteria:

1. Age<18
2. Individuals not belonging to the 3 cohorts of interest listed in the inclusion criteria.
3. Those who are not able to understand written English will be excluded, indeed by the design and methodology of the study, as the study invite and all other information provided is in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Doctors, nurses and other healthcares ≥ 18 years of age in direct contact with patients potentially infected with COVID-19 (n = minimum 800)
  Healthcare /NHS Administrative staff who are working in the hospital, but not directly in contact with patients potentially infected with COVID-19 (minimum n= 125) (internal control)
  Non-healthcare/non-NHS academic staff who are not working in the environment where patient exposure is expected (minimum n=125) (population control)
Sampling Method: Non-Probability Sample
Enrollment: 1721 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Presence of anxiety at baseline | baseline
  Symptoms of anxiety will be investigated using the 7-item Generalised Anxiety Disorder (GAD- 7) Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
  Higher score corresponding to more severe degree of anxiety.
Presence of depression at baseline | baseline
  Symptoms of depression will be investigated using the 9- item Patient Health Questionnaire (PHQ-9).
  Min score of severity: 0-4 none, 20-27 severe. Higher score corresponding to more severe degree of depression
Proportion of those who report a combined outcome of presence of anxiety or depression at the baseline as determined by screening questionnaires used. | baseline
  Anxiety will be investigated by 7-item Generalised Anxiety Disorder and depression will be investigated by 9-item patient health questionnaire. Presence of either one of those or both will be taken as the combined outcome.
  For anxiety, 7-item Generalized anxiety disorder score (GAD- 7) Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
  Higher score corresponding to more severe degree of anxiety. For depression, the 9- item Patient Health Questionnaire (PHQ-9). Min score of severity: 0-4 none, 20-27 severe. Higher score corresponding to more severe degree of depression
  Higher score corresponding to more severe degree of anxiety.
Change in proportion of who report a combined outcome of either presence of anxiety or depression from baseline to the end of study | 4 months
  Anxiety will be investigated by 7-item Generalised Anxiety Disorder and depression will be investigated by 9-item patient health questionnaire. Presence of either one of those or both will be taken as the combined outcome.
  For anxiety, 7-item Generalized anxiety disorder score (GAD- 7) Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
  Higher score corresponding to more severe degree of anxiety. For depression, the 9- item Patient Health Questionnaire (PHQ-9). Min score of severity: 0-4 none, 20-27 severe. Higher score corresponding to more severe degree of depression
Change in the proportion of those who report signs and symptoms or evidence consistent with probable diagnosis of COVID-19 from baseline to the end of study | 4 months
  Self reported, assessed based on the questions regarding the presence of symptoms with presence of either self reported positive test, or self-isolation of 7 or more days.

SECONDARY OUTCOMES:
Change in prevalence of anxiety from baseline | 4 months
  Symptoms of anxiety will be investigated using the 7-item Generalised Anxiety Disorder (GAD- 7) Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
  Higher score corresponding to more severe degree of anxiety.
Change in prevalence of depression from baseline | 4 months followup
  Symptoms of depression will be investigated using the 9- item Patient Health Questionnaire (PHQ-9).
  Min score of severity: 0-4 none, 20-27 severe. Higher score corresponding to more severe degree of depression
Prevalence of sleep-related issues at baseline | At baseline
  This is based on questions derived from the Insomnia Severity Index Total score categories: 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Change in prevalence of sleep-related issues from baseline | 4-month follow-up
  Insomnia Severity Index
  Total score categories: 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Prevalence of a combined outcome of presence of anyone of anxiety, depression or sleep related issues at baseline. | baseline
  Symptoms of depression will be investigated using the 9- item Patient Health Questionnaire (PHQ-9).
  Min score of severity: 0-4 none, 20-27 severe. Higher score corresponding to more severe degree of depression
  Symptoms of anxiety will be investigated using the 7-item Generalised Anxiety Disorder (GAD- 7) Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
  Higher score corresponding to more severe degree of anxiety.
  Total score categories: 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Proportion of those with low mental wellbeing at baseline | baseline
  This is based on questions derived from the Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS). Scores of 7-17 represent probable depression or anxiety; Scores of 18-20 suggest possible depression or anxiety.
Change in proportion of those with low mental wellbeing from baseline to the end of study. | 4-month follow-up
  Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS). Scores of 7-17 represent probable depression or anxiety; Scores of 18-20 suggest possible depression or anxiety
Prevalence of those who report concern related to work-place practices. | At baseline
  Self-reported measures through responses to direct questions relevant to work-related practices in the survey
Change in the prevalence from baseline of those who report concern related to work-place practices. | 6-week
  Self-reported measures through responses to direct questions relevant to work-related practices in the survey
Change in the prevalence from baseline of those who report concern related to work-place practices. | 4 months
  Self-reported measures through responses to direct questions relevant to work-related practices in the survey
Change in behavioural habits, such as smoking and alcohol intake from baseline to the end of study | 4-month follow-up
  Self-reported measures through responses to survey questions
Proportion of those who report signs and symptoms or evidence consistent with probable diagnosis of COVID-19 | Baseline
  Self reported, based on the presence of symptoms with either self reported positive test, or self-isolation of 7 or more days.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gupta, MD, PhD, Principal Investigator — Queen Mary University London
Locations (1):
- Ajay K Gupta, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Collett G, Kotecha A, Gupta A. Burnout and Depression Among UK-Based Healthcare Professionals: Insights From a 3-Year Prospective Cohort Study Regarding Potential Mitigation Strategies. J Occup Environ Med. 2025 Jul 1;67(7):477-482. doi: 10.1097/JOM.0000000000003364. Epub 2025 Feb 21. PMID 40063847
- [Derived] Siddiqui I, Gupta J, Collett G, McIntosh I, Komodromos C, Godec T, Ng S, Maniero C, Antoniou S, Khan R, Kapil V, Khanji MY, Gupta AK; CoPE-HCP clinical investigators. Perceived workplace support and mental health, well-being and burnout among health care professionals during the COVID-19 pandemic: a cohort analysis. CMAJ Open. 2023 Feb 28;11(1):E191-E200. doi: 10.9778/cmajo.20220191. Print 2023 Jan-Feb. PMID 36854456
- [Derived] Khanji MY, Collett G, Godec T, Maniero C, Ng SM, Siddiqui I, Gupta J, Kapil V, Gupta A. Improved lifestyle is associated with improved depression, anxiety and well-being over time in UK healthcare professionals during the COVID-19 pandemic: insights from the CoPE-HCP cohort study. Gen Psychiatr. 2023 Jan 20;36(1):e100908. doi: 10.1136/gpsych-2022-100908. eCollection 2023. PMID 36751400
- [Derived] Khanji MY, Maniero C, Ng S, Siddiqui I, Gupta J, Crosby L, Antoniou S, Khan R, Kapil V, Gupta A. Early and Mid-Term Implications of the COVID-19 Pandemic on the Physical, Behavioral and Mental Health of Healthcare Professionals: The CoPE-HCP Study Protocol. Front Psychol. 2021 Feb 2;12:616280. doi: 10.3389/fpsyg.2021.616280. eCollection 2021. PMID 33603701